CLINICAL TRIAL: NCT02428244
Title: Let's STOP Now Trial: Smoking in Trauma Orthopaedic Patients. A Prospective Randomized Trial
Brief Title: Let's STOP Now Trial: Smoking in Trauma Orthopaedic Patients
Acronym: STOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Maryland Department of Health and Mental Hygiene (Other Government)
Responsible Party: Principal Investigator, Robert O'Toole, Division Chief, Orthopaedic Trauma, Department of Orthopaedics, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HP-00061647
Record Dates: First submitted 2014-11-12; First posted 2015-04-28 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Smoking, Tobacco; Fractures, Bone
Keywords: Smoking; Cessation; Trauma; Fracture; Complications
MeSH Terms: conditions — Tobacco Smoking; Fractures, Bone; Smoking; Wounds and Injuries | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1, Control (No Intervention): Standard of care intervention: All patients at the University as a standard of care receive informational materials about smoking cessation. They are referred to the patient resource center at our institution. Patients will be provided this, also they will be provided with a smoking cessation Quitline Brochure
- Standard of care + brief counseling (Experimental): Patients who are randomized into this arm will receive the standard of care (outlined above). Additionally, patients will also receive a smoking education/counseling session. Patients will receive 10-30 minutes of guided discussion regarding the risks and benefits with regards to smoking and the healing of their traumatic injuries. The smoking educators, who will be trained in accordance with the guidelines provided by MdQuit.org will utilize motivational interviewing techniques to enhance interest in quitting. Patients will receive a description of the quitline, and the quitlined will be the recommended resource. If patients elect to enroll in the quitline, they will be consented using the standardized quitline protocols.
  Interventions: Behavioral: Motivational Interviewing
- Standard of care + counseling/follow-up (Experimental): Patients who are randomized into this arm will receive the same intervention as patients in Arm 2, except when patients arrive for their follow-up, the smoking educator will "check-in" with their progress for approximately 5 minutes. The techniques utilized during this check-in visit will include repetition of previously described motivational interviewing, at this point patients who elect to be referred to the quitline will be given this opportunity.
  Interventions: Behavioral: Motivational Interviewing + Follow-up

INTERVENTIONS:
Behavioral: Motivational Interviewing — Motivational Interviewing coupled with education will be provided to help participants understand the risks associated with smoking and their fracture care. They will be referred to the quitline.
  Arms: Standard of care + brief counseling
Behavioral: Motivational Interviewing + Follow-up — Motivational Interviewing coupled with education will be provided to help participants understand the risks associated with smoking and their fracture care. They will be referred to the quitline.
  In this intervention, the participants will receive additional motivational interviewing sessions at 2 weeks, 6 weeks, 3 months and 6 months.
  Arms: Standard of care + counseling/follow-up

SUMMARY:
It is well known that smoking has deleterious effects to fracture/broken bone outcomes. Complications associated with smoking can be mitigated by smoking cessation. Initiating smoking cessation programs while patients are in the inpatient hospital setting has shown to be an opportune time to enroll patients in a smoking cessation program. The goal of this study is to determine if inpatient smoking counseling with/without follow-up is superior to the standard smoking cessation information associated with admission to a hospital facility.

DETAILED DESCRIPTION:
Patients who elect to be enrolled in the study will receive an initial enrollment survey (attached, Initial Survey) and baseline exhaled carbon monoxide (see below) and be in one of three arms. The arms in brief include (1) standard of care with research follow-up (as mentioned in the below protocol, control arm), (2) standard of care + a 10-30 minute discussion while an inpatient in the hospital regarding the negative effects of smoking with regards to their traumatic injury with research follow-up, and finally (3) standard of care + a 10-30 minute discussion while an inpatient in the hospital regarding the negative effects of smoking with regards to their traumatic injury with research follow-up and follow-up with the investigators smoking educator.

Participants in arms 2 and 3 will receive their education session at the time of enrollment. Research follow-up (as outlined below) will be conducted at the time of normal clinic visits (to avoid unnecessary visits by the patient for the purposes of research), or over the phone if the patient is unable to make the appointment. Arm 3, which includes 'follow-up with the investigators smoking educator' will receive follow-up with the smoking educator at the time of their research follow-up, eliminating the need for additional visits.

Descriptions of arms:

Arm 1, Control: Standard of care intervention: All patients at the University as a standard of care receive informational materials about smoking cessation. They are referred to the patient resource center. The brochure/document that patients are given which details the resources available is standardized. Patients will be provided this, also they will be provided with a Quitline Brochure.

Arm 2, Standard of care + brief counseling: Patients who are randomized into this arm will receive the standard of care (outlined above). Additionally, patients will also receive a smoking education/counseling session. Patients will receive 10-30 minutes of guided discussion regarding the risks and benefits with regards to smoking and the healing of their traumatic injuries. The smoking educators, who will be trained in accordance with the guidelines provided by MdQuit.org will utilize motivational interviewing techniques to enhance interest in quitting. Patients will receive a description of the quitline, and the quitlined will be the recommended resource. If patients elect to enroll in the quitline, they will be consented using the standardized quitline consent/referral form .

Arm 2, Standard of care + brief counseling + extended follow-up: Patients who are randomized into this arm will receive the same intervention as patients in Arm 2, except when patients arrive for their follow-up, the smoking educator will "check-in" with their progress for approximately 5 minutes. The techniques utilized during this check-in visit will include repetition of previously described motivational interviewing, at this point patients who elect to be referred to the quitline will be given this opportunity.

Research follow-up: All participants in the study will receive follow-up at approximate intervals of 2 weeks, 6 weeks, 3 months, and 6 months. These time points were selected as they most closely align with clinical follow-up. Patients will receive their research follow-up at the time of their scheduled clinical encounters, to prevent the participant from having to make additional visits. If the participants are unable to make the visits, or their clinical follow-up is not within 1 week of expected timepoint, follow-up will be attempted via phone. All patients during their follow-up visit will receive the follow-up survey. This survey includes the primary outcome, which is self-reported 7-day abstinence from smoking. Additionally, patients exhaled carbon monoxide level will be measured at these intervals using a standard carbon monoxide meter that is frequently used in research (Pico+ Smokerylyzer, Bedfont Scientific, Haddonfield, NJ, USA). A reference of 8ppm will be utilized to determine abstinence. Otherwise, no other deviation from the standard of care will occur. In the event that patients are unable to follow-up at these schedule intervals, attempt will be made to contact the participants over the phone to perform the survey, and if possible, arrange a visit to perform the exhaled carbon monoxide metering.

At all time points patients will have the ability to receive the informational materials or referral to the quitline that had been received at the time of enrollment.

Conclusion of the patients involvement in the study will occur at their 6-month follow-up visit.

Referral to the quitline will be recorded. Successful referral will be defined as patients who sign the referral form. As part of the standard usage of the quitline and permission of the participant, the quitline will notify us the participants progress via their fax-to-assist program. Information including number of phone calls, services utilized (nicotine patches, text messaging, etc.) will be provided, in addition to self-reported abstinence at 6 months. This will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Active smoker (defined as having smoked some days or every day within the last six months
2. Identifying with having some interest in quitting smoking
3. Sustained an orthopaedic injury requiring surgery
4. Age 18 or older
5. Following up at our institution
6. Ability to consent within 3 weeks of first operative intervention
7. Anticipated acute hospital discharge before first follow-up (2-3 weeks)
8. Cognitive ability to consent

Exclusion Criteria:

1. Age 80 or older
2. Cognitive Inability to consent
3. Having previously utilized the Maryland Quitline
4. Not having a reliable phone line (i.e. conventional land line or cell phone)
5. Inability or refusal to follow-up at the designated follow-up time points

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2014-11; Primary Completion 2018-10-24 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Change in 7-day abstinence point prevalence at 2 weeks | 2 weeks
  Self-reported 7-day abstinence from smoking at 2 weeks
Change in 7-day abstinence point prevalence at 6 weeks | 6 weeks
  Self-reported 7-day abstinence from smoking at 6 weeks
Change in 7-day abstinence point prevalence at 3 months | 3 months
  Self-reported 7-day abstinence from smoking at 3 months
Change in 7-day abstinence point prevalence at 6 months | 6 months
  Self-reported 7-day abstinence from smoking at 6 months

SECONDARY OUTCOMES:
Change in Use of the Quitline at 2 weeks | 2 weeks
  Successful referral and use of quitline at 2 weeks
Change in Use of the Quitline at 6 weeks | 6 weeks
  Successful referral and use of quitline at 6 weeks
Change in Use of the Quitline at 3 months | 3 months
  Successful referral and use of quitline at 3 months
Change in Use of the Quitline at 6 months | 6 months
  Successful referral and use of quitline at 6 months
Change in Exhaled Carbon Monoxide at 2 weeks | 2 week
  Abstinence defined as 8-ppm exhaled carbon monoxide at 2 weeks
Change in Exhaled Carbon Monoxide at 6 weeks | 6 weeks
  Abstinence defined as 8-ppm exhaled carbon monoxide at 6 weeks
Change in Exhaled Carbon Monoxide at 3 months | 3 months
  Abstinence defined as 8-ppm exhaled carbon monoxide at 3 months
Change in Exhaled Carbon Monoxide at 6 months | 6 months
  Abstinence defined as 8-ppm exhaled carbon monoxide at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Matuszewski, MD, Study Director — University of Maryland, Department of Orthopaedics
Locations (1):
- University of Maryland, Shock Trauma Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Scolaro JA, Schenker ML, Yannascoli S, Baldwin K, Mehta S, Ahn J. Cigarette smoking increases complications following fracture: a systematic review. J Bone Joint Surg Am. 2014 Apr 16;96(8):674-81. doi: 10.2106/JBJS.M.00081. PMID 24740664
- [Background] Stephens BF, Murphy A, Mihalko WM. The effects of nutritional deficiencies, smoking, and systemic disease on orthopaedic outcomes. J Bone Joint Surg Am. 2013 Dec 4;95(23):2152-7. doi: 10.2106/00004623-201312040-00010. No abstract available. PMID 24449933
- [Background] Lee JJ, Patel R, Biermann JS, Dougherty PJ. The musculoskeletal effects of cigarette smoking. J Bone Joint Surg Am. 2013 May 1;95(9):850-9. doi: 10.2106/JBJS.L.00375. PMID 23636193
- [Background] Nasell H, Ottosson C, Tornqvist H, Linde J, Ponzer S. The impact of smoking on complications after operatively treated ankle fractures--a follow-up study of 906 patients. J Orthop Trauma. 2011 Dec;25(12):748-55. doi: 10.1097/BOT.0b013e318213f217. PMID 21886001
- [Background] Rabe GL, Wellmann J, Bagos P, Busch MA, Hense HW, Spies C, Weiss-Gerlach E, McCarthy W, Gareca Arizaga MJ, Neuner B. Efficacy of emergency department-initiated tobacco control--systematic review and meta-analysis of randomized controlled trials. Nicotine Tob Res. 2013 Mar;15(3):643-55. doi: 10.1093/ntr/nts212. Epub 2012 Sep 27. PMID 23024250
- [Background] Dohnke B, Ziemann C, Will KE, Weiss-Gerlach E, Spies CD. Do hospital treatments represent a 'teachable moment' for quitting smoking? A study from a stage-theoretical perspective. Psychol Health. 2012;27(11):1291-307. doi: 10.1080/08870446.2012.672649. Epub 2012 Apr 4. PMID 22472171
- [Background] Fu SS, McFall M, Saxon AJ, Beckham JC, Carmody TP, Baker DG, Joseph AM. Post-traumatic stress disorder and smoking: a systematic review. Nicotine Tob Res. 2007 Nov;9(11):1071-84. doi: 10.1080/14622200701488418. PMID 17978982
- [Background] Spencer L, Pagell F, Hallion ME, Adams TB. Applying the transtheoretical model to tobacco cessation and prevention: a review of literature. Am J Health Promot. 2002 Sep-Oct;17(1):7-71. doi: 10.4278/0890-1171-17.1.7. PMID 12271754
- [Background] DiClemente CC, Prochaska JO, Fairhurst SK, Velicer WF, Velasquez MM, Rossi JS. The process of smoking cessation: an analysis of precontemplation, contemplation, and preparation stages of change. J Consult Clin Psychol. 1991 Apr;59(2):295-304. doi: 10.1037//0022-006x.59.2.295. PMID 2030191
- [Background] DiClemente CC, Delahanty JC, Fiedler RM. The journey to the end of smoking: A personal and population perspective. Am J Prev Med. 2010 Mar;38(3 Suppl):S418-28. doi: 10.1016/j.amepre.2009.12.010. PMID 20176317
- [Background] Hajek P. Individual differences in difficulty quitting smoking. Br J Addict. 1991 May;86(5):555-8. doi: 10.1111/j.1360-0443.1991.tb01807.x. PMID 1859918
- [Background] Blumenthal DS. Barriers to the provision of smoking cessation services reported by clinicians in underserved communities. J Am Board Fam Med. 2007 May-Jun;20(3):272-9. doi: 10.3122/jabfm.2007.03.060115. PMID 17478660
- [Background] Risser NL, Belcher DW. Adding spirometry, carbon monoxide, and pulmonary symptom results to smoking cessation counseling: a randomized trial. J Gen Intern Med. 1990 Jan-Feb;5(1):16-22. doi: 10.1007/BF02602303. PMID 2405112
- [Background] Chen CC, Chang CH, Tsai YC, Tseng CW, Tu ML, Wang CC, Lin MC, Liu SF. Utilizing exhaled carbon monoxide measurement with self-declared smoking cessation: enhancing abstinence effectiveness in Taiwanese outpatients. Clin Respir J. 2015 Jan;9(1):7-13. doi: 10.1111/crj.12096. Epub 2014 Jan 17. PMID 24345098
- [Background] Brugger OE, Frei M, Sendi P, Reichart PA, Ramseier CA, Bornstein MM. Assessment of smoking behaviour in a dental setting: a 1-year follow-up study using self-reported questionnaire data and exhaled carbon monoxide levels. Clin Oral Investig. 2014 Apr;18(3):909-15. doi: 10.1007/s00784-013-1036-x. Epub 2013 Jul 20. PMID 23873321
- [Background] Javors MA, Hatch JP, Lamb RJ. Cut-off levels for breath carbon monoxide as a marker for cigarette smoking. Addiction. 2005 Feb;100(2):159-67. doi: 10.1111/j.1360-0443.2004.00957.x. PMID 15679745
- [Background] Rigotti NA, Regan S, Levy DE, Japuntich S, Chang Y, Park ER, Viana JC, Kelley JH, Reyen M, Singer DE. Sustained care intervention and postdischarge smoking cessation among hospitalized adults: a randomized clinical trial. JAMA. 2014 Aug 20;312(7):719-28. doi: 10.1001/jama.2014.9237. PMID 25138333